CLINICAL TRIAL: NCT00320229
Title: Half-Dose Intracoronary Abciximab Bolus Improves the Mortality Outcome Compared to Standard Intravenous Regimen
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Sanitaria Ospedaliera (Other)
Collaborators: Cardiologia 2 - Emodinamica - Ospedale Maggiore, Novara, Italy (Unknown)
Other Study IDs: ABCX-LD
Record Dates: First submitted 2006-04-18; First posted 2006-05-03 (Estimated); Last update posted 2006-05-16 (Estimated); Status verified 2006-01

CONDITIONS: Coronary Disease; Myocardial Infarction
Keywords: angioplasty; stent; abciximab; Platelet Glycoprotein GPIIb-IIIa Complex; myocardial infarction
MeSH Terms: conditions — Coronary Disease; Myocardial Infarction | interventions — Abciximab

INTERVENTIONS:
Drug: abciximab

SUMMARY:
The aim of our study was to demonstrate that, during a percutaneous coronary intervention, even smaller amounts of abciximab than standard dose, injected locally, could achieve a rapid thrombus resolution and clinical improvement without concomitant differences in hemorrhagic complications

DETAILED DESCRIPTION:
Patients both with acute myocardial infarction and unstable angina are prone to extensive intracoronary thrombosis, leading to acute deterioration during percutaneous coronary intervention or thrombosis of the device despite therapy. Intracoronary use of abciximab has reported favourable results. We randomly assigned 84 patients to intracoronary half abciximab bolus (group A) and to standard regimen (group B).

ELIGIBILITY:
Inclusion Criteria:

* presenting with unstable angina
* presenting with acute myocardial infarction
* eligibility for percutaneous coronary intervention

Exclusion Criteria:

* presenting with cardiogenic shock

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84
Dates: Start 2004-12; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: Mara Sansa, Principal Investigator — Chief Interventional Cardiology - Ospedale Maggiore - Novara - Italy
Locations (1):
- Cardiologia 2 - Emodinamica - Ospedale Maggiore, Novara, Italy